CLINICAL TRIAL: NCT02225808
Title: Neural Mechanisms of Cognitive-Behavioral Therapy for Anxiety in Children With Autism Spectrum Disorder: A Pilot Study
Brief Title: Neural Mechanisms of CBT for Anxiety in Autism (Open Pilot Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1211011144
Record Dates: First submitted 2014-08-19; First posted 2014-08-26 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Autism; Autism Spectrum Disorder; Anxiety
Keywords: CBT; autism; anxiety; treatment; fMRI
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CBT for anxiety in autism (Experimental): Cognitive-behavioral therapy (CBT) teaches skills for coping with anxiety and consist of 12 weekly sessions. CBT is conducted with child and parent.
  Interventions: Behavioral: CBT for anxiety in autism

INTERVENTIONS:
Behavioral: CBT for anxiety in autism

SUMMARY:
This is an open, pilot study of neural mechanisms of cognitive-behavioral therapy for anxiety in children with high-functioning autism spectrum disorder (ASD). In addition to the core symptoms, approximately forty percent of children with ASD exhibit clinically significant levels of anxiety. Cognitive-Behavioral Therapy (CBT) is a promising treatment for anxiety in children with high-functioning ASD, but the neural mechanisms of this treatment have not been studied. CBT teaches emotion regulation skills such as cognitive reappraisal, followed by behavioral exposure to anxiety-provoking situations. The investigators propose to investigate the neural mechanisms of CBT for anxiety by evaluating fMRI indices of socioemotional functioning before and after treatment in children, ages 8 to 14, with high-functioning ASD. Dysfunction of the amygdala and its connectivity with prefrontal cortex has been implicated in co-occurring ASD and anxiety. In the investigators research, compared to typically developing controls, children with ASD have shown lower activation in several regions of prefrontal cortex and a lack of down-regulation in the amygdala during a task of emotion regulation. Based on these observations, the investigators propose that a positive response to CBT for anxiety in children with ASD will be associated with increased activation of several regions in the prefrontal cortex as well as increased functional connectivity between prefrontal regions the amygdala during the task of emotion regulation. The primary aim of this pilot study is to examine the effects of CBT on the neural basis of anxiety in ASD by collecting fMRI data during emotion regulation, face perception, and rest before and after treatment. The investigators hypothesize that CBT will increase prefrontal activity, decrease amygdala reactivity, and enhance amygdala-prefrontal functional connectivity during emotion regulation. The investigators also hypothesize that CBT will decrease amygdala reactivity during perception of emotional faces. Additional analyses will be conducted to explore change in resting-state functional connectivity before and after CBT for anxiety in children with ASD.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, ages 8 to 14 inclusive.
2. DSM-V diagnosis of autism spectrum disorder.
3. DSM-V diagnosis of generalized anxiety disorder, separation anxiety disorder, or social phobia.
4. Score > 19 on the 20 Item Anxiety scale of the Child and Adolescent Symptom Inventory.
5. Full Scale IQ and Verbal IQ > 70.
6. Unmedicated or on stable medication for irritability, ADHD, anxiety, or depression for at least 6 weeks, with no planned changes for duration of study.

7. Subjects will be free of metal medical implants, and will have a body weight of less than 250 lbs. and no claustrophobia. [These are necessitated by the safety requirements of the fMRI.]

8. Child is an English speaker.

9. Child is able to meet fMRI data quality requirements at baseline [to enable pre- to post-treatment comparison.]

Exclusion Criteria:

1. Presence of a known serious medical condition in the child (based on medical history or parent report) that would interfere with child and parent's ability to participate in the study.
2. Presence of a current psychiatric diagnosis in the child that would require alternative treatment (based on assessment by experienced study clinician).
3. Previous treatment with four or more sessions of CBT for anxiety. -

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2014-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
functional magnetic resonance imaging (fMRI) | baseline (week 0)
  fMRI scanning with tasks of emotion regulation and social perception
functional magnetic resonance imaging (fMRI) | endpoint (week 12)
  fMRI scanning with tasks of emotion regulation and social perception

SECONDARY OUTCOMES:
Multidimensional anxiety scale for children (MASC) | baseline (week 0)
  parent rating of child anxiety
Multidimensional anxiety scale for children (MASC) | endpoint (week 12)
  parent rating of child anxiety
Pediatric Anxiety Rating Scale (PARS) | baseline (week 0)
  clinician rating of anxiety based on an interview with parent and child
Pediatric Anxiety Rating Scale (PARS) | endpoint (week 12)
  clinician rating of anxiety based on an interview with parent and child

CONTACTS AND LOCATIONS:
Overall Officials: Denis Sukhodolsky, Ph.D., Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, Child Study Center, New Haven, Connecticut, United States

REFERENCES:
- [Background] Sukhodolsky DG, Bloch MH, Panza KE, Reichow B. Cognitive-behavioral therapy for anxiety in children with high-functioning autism: a meta-analysis. Pediatrics. 2013 Nov;132(5):e1341-50. doi: 10.1542/peds.2013-1193. Epub 2013 Oct 28. PMID 24167175
- [Background] Sukhodolsky DG, Scahill L, Gadow KD, Arnold LE, Aman MG, McDougle CJ, McCracken JT, Tierney E, Williams White S, Lecavalier L, Vitiello B. Parent-rated anxiety symptoms in children with pervasive developmental disorders: frequency and association with core autism symptoms and cognitive functioning. J Abnorm Child Psychol. 2008 Jan;36(1):117-28. doi: 10.1007/s10802-007-9165-9. Epub 2007 Aug 3. PMID 17674186